CLINICAL TRIAL: NCT06048913
Title: Nimotuzumab Combined With Concurrent Chemoradiotherapy for Locally Advanced Treatment Esophageal Cancer in Old Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GXL-002
Record Dates: First submitted 2023-03-16; First posted 2023-09-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Carcinoma
Keywords: Nimotuzumab; Concurrent chemoradiotherapy; Locally advanced esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — nimotuzumab; S 1 (combination); Drug Therapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab combined with concurrent chemoradiotherapy (Experimental): Treatment options Nimotuzumab （400mg plus normal saline 250ml intravenous infusion for not less than 60 minutes. Starting from week 1 of radiotherapy, 1 dose of the same dose each time for a total of 6 doses）combined with chemoradiotherapy (Oral chemotherapy with the tigio regimen is given on days 1 to 2 of radiotherapy, with the drug dose calculated based on body surface area, and the oral S-1 course from Monday to Friday is synchronized with radiation therapy) for the treatment of locally advanced elderly esophageal cancer patients, in which the S-1 regimen with good clinical tolerability was selected for chemotherapy to evaluate the short-term efficacy and toxic side effects
  Interventions: Drug: Nimotuzumab; Drug: S-1; Radiation: Concurrent radiation therapy

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 400mg plus normal saline 250ml intravenous infusion for not less than 60 minutes. Starting from week 1 of radiotherapy, 1 dose of the same dose each time for a total of 6 doses. The use of nimotuzumab is not interrupted due to interruption of radiotherapy during the administration until the end of radiotherapy.
  Other Names: taixinsheng
Drug: S-1 — Oral chemotherapy with the S-1 regimen is given on days 1 to 2 of radiotherapy, with the drug dose calculated based on body surface area, and the oral S-1 course from Monday to Friday is synchronized with radiation therapy.
  Other Names: chemotherapy
Radiation: Concurrent radiation therapy — Outline the target area layer by layer on the enhanced CT image, PGTV, PTV. The endangered organs are delineated layer by layer on the cross-section, and extended 0.3cm to form a corresponding plan to endanger the organs. The reverse intensity modulated radiotherapy plan was designed on the Monaco treatment plan system, with a prescribing dose of 56Gy/30F for PTV and 60Gy/30F for pGTV, and the target dose distribution and organ exposure dose were evaluated layer by layer on a cross-sectional surface, and combined with dose-to-volume histogram (DVH) evaluation and optimal treatment plan, the maximum dose of radiation in the spinal cord < 40 Gy and lung V20<30%. After the treatment plan is confirmed, the dose is verified on the treatment machine, and the treatment plan is executed after it is accurate. govern
  Other Names: Chemoradiotherapy

SUMMARY:
The research subjects of this project are mainly aimed at patients with locally advanced esophageal cancer who cannot be treated surgically, in nimotuzumab 3 months after the end of concurrent chemoradiotherapy, RECIST is pressed as based on physical examination and esophageal barium dialysis or esophageal contrast-enhanced CT Criteria assessed short-term and long-term efficacy separately. By detecting the expression of EGFR in patients with locally advanced esophageal cancer, the relationship between the efficacy of EGFR monoclonal antibody therapy and the long-term prognosis of patients was evaluated. Evaluation of safety, toxicity and side effects during treatment and in the near and long term.

DETAILED DESCRIPTION:
It is expected that 52 patients will be enrolled, and patients who meet the enrollment criteria will undergo esophagoscopy, esophageal barium meal examination, chest contrast-enhanced CT, abdominal ultrasound, electrocardiogram, blood routine, whole body bone scan, liver and kidney function and other examinations before treatment, and esophageal ultrasound if necessary. Patients who received esophageal ultrasound were staged by esophageal ultrasound results, and those without esophageal ultrasound were mainly staged according to the cervical chest and epigastric contrast CT and esophageal barium plates, and clinical staging was performed according to the 2002 AJCC staging standard. After the combination of nimotuzumab and concurrent chemoradiotherapy, adverse reactions and efficacy evaluation were observed. The expected result is that the local control rate of EGFR monoclonal antibody combined with chemoradiotherapy is improved in patients with locally advanced elderly esophageal squamous cell carcinoma, and there is no significant increase in adverse reactions, and serological indicators such as EGFR can be used as prognostic indicators for esophageal malignancy and have certain guiding significance for treatment. EGFR monoclonal antibody can be used in locally advanced elderly esophageal cancer patients who cannot tolerate chemotherapy, with good short-term efficacy and tolerable toxic side effects, which further provides reference value for clinical guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage II-IVB according to AJCC (8th edition, 2018) (IVB included metastasis to the celiac trunk or supraclavicular lymph nodes only) who are not suitable for or refuse surgery can tolerate concurrent chemoradiotherapy and targeted therapy;
2. The pathological type is esophageal squamous cell carcinoma;
3. Eastern Cooperative Oncology Group performance status of 0-1, age ≥ 75 years old;
4. No serious comorbidities, such as severe obstructive emphysema, hypertension, coronary heart disease, diabetes and psychiatric history, etc., and no other malignant tumors;
5. All patients had not received EGFR-targeted therapy, immunotherapy, and chemoradiotherapy;
6. Expected survival time ≥ 12 weeks.

Exclusion criteria

Patients who meet any of the following criteria will be excluded from this trial:

1. Received EGFR monoclonal antibody or EGFR-TKI within six months;
2. Participated in other interventional clinical trials within 30 days before screening;
3. Patients with serious concurrent diseases, such as heart failure, high-risk uncontrollable arrhythmias, severe myocardial infarction, refractory hypertension, renal failure (CKD-4 and above), thyroid dysfunction, mental illness, diabetes, severe chronic diarrhea (more than 7 bowel movements per day), or patients who are considered unsuitable to participate in this clinical study by the researchers;
4. Patients with brain metastases with symptoms or symptom control time of less than 3 months;
5. Having a history of other malignant tumors (except for cured cervical carcinoma in situ or basal cell carcinoma of the skin and other malignant tumors that have been cured for more than 5 years);
6. The presence of active infection or active infectious disease;
7. Patients with multi-segment esophageal malignant tumors or signs of esophageal fistula or perforation;
8. Patients whose tumors have invaded important blood vessels as shown by imaging or who are judged by the researchers to be very likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study;
9. Those who are allergic to the drugs or their ingredients used in this program;
10. Peripheral neuropathy or hearing loss of grade 2 or higher according to the criteria of Common Terminology for Adverse Events (NCI CTCAE V5.0);
11. Pregnant or breastfeeding women;
12. Patients with a history of psychotropic drug abuse and unable to quit or patients with mental disorders;
13. Those who are considered unsuitable to participate in this study by the researcher;
14. Those who are unwilling to participate in this study or unable to sign the informed consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | up to 3 years
  Progression-free survival was measured from the treatment initiation to either tumor progression (in any form) or death from any cause

SECONDARY OUTCOMES:
complete response，CR | through study completion, an average of 18 month
  After treatment, the lesion completely disappears, or all symptoms and signs of the unmeasurable lesion completely disappear, and the lesion completely disappears in X-ray and bone imaging examinations for bone metastasis, lasting for at least 4 weeks
partial response，PR | through study completion, an average of 18 month
  The sum of the maximum diameters of the target lesion decreases by more than 30% and lasts for more than 4 weeks.
no response，NR | through study completion, an average of 18 month
  At the end of radiotherapy, there is residual tumor or no significant improvement in the lesion, but there are still significant filling defects and worsening of niche or stenosis
Overall survival | 3-year
  Overall survival was defined as the time from the treatment initiation to death from any cause
Toxic side reactions | through study completion, an average of 18 month
  The US Toxicity Evaluation Standard (CTC3. O) is divided into O~4 grades, and the evaluation of acute radiation reactions adopts RTOG/EROTC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin GE, PhD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT06048913/Prot_000.pdf
  • Informed Consent Form (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT06048913/ICF_001.pdf